CLINICAL TRIAL: NCT00002367
Title: An Open-Label, Non-Comparative Study of Saquinavir-SGC in Combination With Zidovudine (AZT) and Lamivudine (3TC) in the Treatment of HIV-1 Infected Patients With No Previous Anti-Retroviral Drug Therapy
Brief Title: A Study of Saquinavir Soft Gelatin Capsules Plus Zidovudine Plus Lamivudine in the Treatment of HIV-1 Infected Patients Who Have Never Taken Anti-HIV Drugs
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 229F; NR15503; M61005
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-08

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; Zidovudine; HIV Protease Inhibitors; Lamivudine; Saquinavir; Reverse Transcriptase Inhibitors; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Saquinavir; Lamivudine; Zidovudine

INTERVENTIONS:
Drug: Saquinavir
Drug: Lamivudine
Drug: Zidovudine

SUMMARY:
To evaluate the efficacy of Saquinavir-SGC combination with Zidovudine and Lamivudine in the treatment of HIV-1 infected patients with no previous anti-retroviral drug therapy.

DETAILED DESCRIPTION:
All enrolled patients will receive the following 3 drug combination: Saquinavir, Zidovudine and Lamivudine. Efficacy and duration of anti-viral response will be evaluated by monitoring of HIV-1 RNA levels. Patients below the detectable limit of 200 copies/ml will be analyzed using the Ultra-direct method with a detection limit of 20 copies/ml. CD4 and CD8 cell counts will also be analyzed.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Plasma HIV-1 RNA titers > 10,000 copies/ml.
* CD4 cell count > 100 cells/mm3.

Exclusion Criteria

Co-existing Condition:

Patients with any of the following conditions will be excluded:

* Any prior anti-retroviral drug therapy.

Prior Medication:

Excluded:

Previous anti-retroviral drug therapy.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - AIDS Healthcare Foundation Labs, Los Angeles, California
  - Urgent Care Ctr / North Broward Hosp District, Fort Lauderdale, Florida